CLINICAL TRIAL: NCT05535218
Title: SURE-02_An Open Label, Single-arm, Phase 2 Study of Perioperative Pembrolizumab Plus Sacituzumab Govitecan, and Bladder-saving Approach, for Patients With Muscle-invasive Bladder Cancer Who Cannot Receive or Refuse Cisplatin-based Chemotherapy
Brief Title: Pembrolizumab-Sacituzumab Govitecan Combination to Treat High-risk, Localized Bladder Cancer
Acronym: SURE-02
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Claudia Guerrieri (Other)
Responsible Party: Sponsor-Investigator, Claudia Guerrieri, Sponsor delegated, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SURE-02; 2024-514569-20-00 (EU CTIS Number)
Record Dates: First submitted 2022-08-09; First posted 2022-09-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Muscle-invasive Urothelial Carcinoma of the Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Other): Single Arm treatment
  Interventions: Drug: Sacituzumab govitecan is a humanized mAb with a hydrolysable linker through which SN-38 is conjugated to the humanized mAb hRS7 IgG1κ to enhance the delivery of SN-38 to Trop-2- expressing tumors, whi

INTERVENTIONS:
Drug: Sacituzumab govitecan is a humanized mAb with a hydrolysable linker through which SN-38 is conjugated to the humanized mAb hRS7 IgG1κ to enhance the delivery of SN-38 to Trop-2- expressing tumors, whi — Neoadjuvant treatment: 7,5mg/kg sacituzumab-govitecan IV, on days 1, 8, of each 21 day cycle; Pembrolizumab will be administered in combination with sacituzumab-govitecan on day 1, every 21 days, at the standard dose of 200 mg intravenously. A total of 4 cycles is planned before surgery.
  After surgery patients will receive additional 13 cycles of pembrolizumab at the standard dose, every 3 weeks, accounting for a total of 17 cycles of perioperative pembrolizumab (neoadjuvant + adjuvant).

SUMMARY:
This is a Phase 2, single-center, open-label, non-randomized study in patients with MIBC who cannot receive or refuse to receive cisplatin-based chemotherapy.

Patients will be consecutively enrolled and treated. All patients enrolled who receive at least 1 cycle of study drug will be included in the primary and secondary endpoint analyses.

DETAILED DESCRIPTION:
The general framework of the study will be as follows:

A TURBT for biopsy, histological characterization, and local staging will be executed first, according to the guidelines. With the aim to improve the sensitivity of CT scan in assessing pelvic lymph-nodes and better assess the local extent of bladder tumor, computed tomography (CT) scan, 18FDG-PET/CT scan, and a pelvic MRI will be done during screening and before the surgical assessment to stage and evaluate response. The same imaging assessments will be performed after the neoadjuvant treatment. Patients with the evidence of no detectable disease after neoadjuvant therapy will also undergo a cystoscopy assessment prior to the reTURBT.

* Eligible patients will receive neoadjuvant treatment: 7.5 mg/kg sacituzumab govitecan IV, on days 1, 8, of each 21 day cycle.
* Pembrolizumab will be administered in combination with sacituzumab govitecan on day 1, every 21 days, at the standard dose of 200 mg intravenously.
* A total of 4 cycles is planned before surgery.
* Patients who achieve a clinical complete response (cCR) will be offered a reTURBT instead of radical cystectomy. Patients not achieving a cCR will undergo a radical cystectomy.
* cCR will be defined as the achievement of ALL the following requirements: no evidence of residual disease (VIRADS 0 score) at MRI, negative cystoscopy, and a biopsy obtained via reTURBT revealing no residual viable cancer.
* Surgery will be planned at the time of study inclusion to be done ideally within 4 weeks of the last dose of study drug, and not later than 12 weeks from the last dose of study drug.
* After surgery patients will receive additional 13 cycles of pembrolizumab at the standard dose, every 3 weeks, accounting for a total of 17 cycles of perioperative pembrolizumab(neoadjuvant + adjuvant).
* After cystectomy or reTURBT, patients will undergo imagingassessments according to EAU guidelines. In patients undergoing reTURBT, cystoscopy assessments will be performed every 4 months for the first 2 years (until study conclusion),then according to investigator judgment.
* At the end of the adjuvant period, patients will enter the follow-up period which will lastuntil 12 months from the last dose of pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects, >18 years of age, able to understand and give written informed consent
2. Histopathologically confirmed urothelial carcinoma. Patients with mixed histologies are required to have a dominant (i.e. 50% at least) transitional cell pattern.
3. Fit and planned for RC (according to local guidelines).
4. ECOG performance status score of 0 or 1.
5. Refusal of unsuitability for standard chemoradiotherapy protocols.
6. Adequate hematologic counts without transfusional or growth factor support within 2 weeks of study drug initiation (Hemoglobin ≥ 9 g/dL, ANC ≥ 1,500/ mm3, and Platelets

   ≥ 100,000/ μL)
7. Adequate hepatic function (Bilirubin ≤ 1.5 IULN, AST and ALT ≤ 2.5 x IULN or ≤ 5 x IULN if known liver metastases and serum albumin >3 g/dl)
8. Creatinine clearance ≥30 mL/min as assessed by the Cockcroft-Gault equation
9. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication, and must not be lactating. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
10. Female subjects of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >2 years
11. Male subjects must agree to use an adequate method of contraception starting with the first dose of study therapy through 3 months after the last dose of study therapy.
12. Clinical stage T2-T3bN0M0 MIBC, assessed by CT + PET/CT + pelvic MRI.
13. The patient accepts to undergo RC.
14. Ineligibility to receive cisplatin-based neoadjuvant chemotherapy based on Galsky's criteria OR refusal to receive neoadjuvant cisplatin-based chemotherapy.

Exclusion Criteria:

1. Have received prior systemic anti-cancer therapy including investigational agents and immunotherapy.
2. Have received prior radiotherapy on the bladder tumor.
3. Have received a partial cystectomy.
4. Refusal to undergo RC.
5. Have received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella,varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
6. Have received any antibiotics within 30 days prior to the first dose of study drug.
7. Are currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigationalagent.
8. Have a known additional malignancy that is progressing or has required active treatment within the past 3 years.
9. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded. Participants with low-risk early stage prostate cancer defined as follows are not excluded; Stage T1c or T2a with a Gleason score ≤ 6 and prostatic-specific antigen (PSA) < 10 ng/mL either treated with definitive intent or untreated in active surveillance that has been stable for the past year prior to study allocation.
10. Have severe hypersensitivity (≥Grade 3) to pembrolizumab or sacituzumab govitecan and/or any of its excipients.
11. Have active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

    Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Have a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
13. Have nephrostomy, central venous catheters, any other types of catheters that could make the patient at higher risk of developing severe infectious complications during treatment with sacituzumab govitecan.
14. Have >=3 risk factors for the development of febrile neutropenia according to the ASCO guidelines (Smith et al, J Clin Oncol. 2015;33:3199-3212). These risk factors are the following: Age >65 years, advanced disease, Previous chemotherapy or radiation therapy, Preexisting neutropenia or bone marrow involvement with tumor, infection, Open woundsor recent surgery, Poor performance status or poor nutritional status, Poor renal function, Liver dysfunction, most notably elevated bilirubin, Cardiovascular disease, Multiple comorbid conditions, HIV infection.
15. Have a history of inflammatory bowel disease, ulcerative colitis, or any other pre-existing inflammatory or autoimmune disease that could make the patient at higher risk of developing severe diarrhea or related complications.
16. Have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Have active cardiac disease, defined as:

    * Myocardial infarction or unstable angina pectoris within 6 months of C1D1
    * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication);
    * history of QT interval prolongation NYHA Class III or greater congestive heart failure or left ventricular ejection fraction of < 40%
18. Have known history of HIV-1/2 infection.
19. Have a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
20. Have other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
21. High dose systemic corticosteroids (≥20 mg of prednisolone or its equivalent) are not allowed within 2 weeks of C1D1.
22. Have received or are currently receiving (within the previous 2 weeks) antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Clinical CR-rate | 36 months
  To assess whether sacituzumab govitecan plus pembrolizumab is an effective perioperative strategy in patients with clinical T2-3bN0M0 MIBC who cannot receive or refuse to receive cisplatin-based chemotherapy.

SECONDARY OUTCOMES:
Pathological response-rate, | Upon completion of the study up to 40 months
  To evaluate the proportion of patients who will be pathological responders.
Bladder-intact event-free survival (BI-EFS); | Up to 6 months
  To evaluate the surgical and medical safety of neoadjuvant combination therapy, as well as of the adjuvant pembrolizumab therapy.
Overall survival | Up to 40 months
  To assess survival outcomes (event-free survival and overall survival), in the total population and in the subgroups according to the pathological response.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Necchi, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Fondazione San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No